CLINICAL TRIAL: NCT01468584
Title: A Phase 3 Study of MP-424 in Combination With Peginterferon Alfa-2b and Ribavirin, in Subjects With Genotype 2 Hepatitis C, Who Did Not Respond to Previous Treatment
Brief Title: Efficacy and Safety of MP-424, Peginterferon Alfa-2b and Ribavirin in Non-responder Genotype 2 Hepatitis C Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G060-A11
Record Dates: First submitted 2011-11-02; First posted 2011-11-09 (Estimated); Results first posted 2014-11-03 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Chronic Hepatitis C
Keywords: Genotype 2
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MP-424 (Experimental)
  Interventions: Drug: MP-424 (generic name:Telaprevir); Drug: Ribavirin; Drug: Peginterferon alfa-2b

INTERVENTIONS:
Drug: MP-424 (generic name:Telaprevir) — 750mg q8h for 12 weeks
Drug: Ribavirin — 400 - 1000 mg/day based on body weight for 24 weeks
Drug: Peginterferon alfa-2b — 1.5mcg/kg/week for 24 weeks

SUMMARY:
This study will evaluate the efficacy and safety of MP-424 with Peginterferon Alfa-2b and Ribavirin (RBV) in patients with genotype 2 hepatitis C, who did not respond to previous treatment.

ELIGIBILITY:
Inclusion Criteria:

* Genotype 2, chronic hepatitis C
* Non-responders (patient who did not respond to previous treatment)
* Able and willing to follow contraception requirements

Exclusion Criteria:

* Cirrhosis of the liver or hepatic failure
* Hepatitis B surface antigen-positive or HIV antibodies-positive
* History of, or concurrent hepatocellular carcinoma
* History of, or concurrent depression, schizophrenia,; or suicide attempt in the past
* Pregnant, lactating, or suspected pregnant patients, or male patients whose female partner is pregnant

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kazuoki Kondo, MD, Study Director — Tanabe Pharma Corporation
Locations (1):
- Toranomon Hospital, Minato-ku, Tokyo, Japan

REFERENCES:
- [Result] Kumada H, Sato K, Takehara T, Nakamuta M, Ishigami M, Chayama K, Toyota J, Suzuki F, Nakayasu Y, Ochi M, Yamada I, Okanoue T. Efficacy of telaprevir-based therapy for difficult-to-treat patients with genotype 2 chronic hepatitis C in Japan. Hepatol Res. 2015 Jul;45(7):745-54. doi: 10.1111/hepr.12416. Epub 2014 Nov 18. PMID 25196718

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MP-424
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MP-424
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Undetectable HCV RNA at 24 Weeks After Completion of Drug Administration (SVR, Sustained Viral Response)
Time Frame: After 24 weeks of follow-up
Measure: Number (95% Confidence Interval); unit: percentage of subjects achieving SVR
Arm/Group | MP-424
Number analyzed (Participants) | 10
percentage of subjects achieving SVR | 50.0 [18.7 to 81.3]

ADVERSE EVENTS:
Arm/Group | MP-424
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MP-424 (N=10)
Nasopharyngitis (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 7
Hyperthyroidism (Endocrine disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Insomnia (Psychiatric disorders) | 1
Headache (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 1
Parosmia (Nervous system disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 1
Generalised erythema (Skin and subcutaneous tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Injection site reaction (General disorders) | 6
Malaise (General disorders) | 4
Pyrexia (General disorders) | 4
Injection site erythema (General disorders) | 3
Chills (General disorders) | 1
Injection site pruritus (General disorders) | 1
Blood bilirubin increased (Investigations) | 5
Blood uric acid increased (Investigations) | 4
Platelet count decreased (Investigations) | 4
White blood cell count decreased (Investigations) | 3
Hyaluronic acid increased (Investigations) | 3
Blood calcium decreased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Blood phosphorus decreased (Investigations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other